CLINICAL TRIAL: NCT06323603
Title: Biomonitoring of Occupationally Populations Exposed to Micro and Nanoplastic
Status: Recruiting | Type: Observational
Sponsor: Ricard Marcos (Other)
Collaborators: Finnish Institute of Occupational Health (Other)
Responsible Party: Sponsor-Investigator, Ricard Marcos, Professor, Universitat Autonoma de Barcelona
Organization: Universitat Autonoma de Barcelona (Other)
Other Study IDs: 3-1
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Occupational Exposure; Genotoxicity; Damage Dna
Keywords: Biomonitoring; Genotoxic damage; Micro and nanoplastic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood, exhaled breath condensate, exfoliated buccal cells, urine and feces
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1. Textile industry workers: Workers from the textile industry, that manufactures non-wovens fibers
  Interventions: Other: Micro and nanoplastic
- 2. Plastic Recycling Workers: Workers involved in recycling and waste management of plastic
  Interventions: Other: Micro and nanoplastic
- 3. Controls: Control group that will match the characteristics of grup 1 and 2

INTERVENTIONS:
Other: Micro and nanoplastic — Biological samples will be obtained to evaluate the different biomarkers selected
  Groups: 1. Textile industry workers; 2. Plastic Recycling Workers

SUMMARY:
The biomonitoring study aims to evaluate genotoxic damage and other parameters of exposure in different occupational exposed populations that work directly with different plastics.

DETAILED DESCRIPTION:
The exponential increase in the production and use of plastic goods translates into a parallel increase of environmental plastic waste that is continuously degraded into micro and nanoplastics (MNPLs). Information on their effects on human health is still preliminary, especially regarding human biomonitoring studies, thus more information is required for risk assessment evaluation.

This observational study aims to evaluate the exposure to MNPLs in human populations occupationally exposed to different types of plastics (fibers and plastic waste). The study will evaluate the effect of exposure to MNPLs (genotoxic and microbiota effects) in different body samples (blood, exfoliated buccal cells, urine,and feces) and also will use those samples to evaluate the presence of MNPLs.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years.
* Healthy subjects defined by the absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, haematology, blood chemistry, and urine analysis.
* Able to participate and willing to give written informed consent and to comply with the study restrictions.
* Have been working at the company for the last 48 months

Exclusion Criteria:

* Workers decline participation
* Legal incapacity or inability to understand or comply with the requirements of the study.
* Any hierarchical subordination to the PI
* Clinically significant findings as determined by medical history taking, physical examination, ECG, and vital signs.
* Submitted to X-ray in the three previous months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study aims to determine whether workers occupationally exposed to different plastics show increased genomic damage, changes in cytokine expression and/ or microbiota. Moreover, the levels of macro/microplastics in different body fluids will be characterized.
  Different European populations dedicated to the recycling of plastics and the production of non-woven textiles will be used, as well as a control group that will match according to the characteristics of the populations.
  At least 50 workers from each of the participating industries will be used to demonstrate a higher exposure MNPLs level and, therefore, an increased health risk.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Characterization of macro and nanoplastics | Up to 1 year
  The characterization of macro and nanoplastics will be done by Raman spectrosmicroscopy and FTIR (From exhaled breath condensate, blood and urine)
Genotoxic evaluation by the Micronucleus assay | Up to 1 year
  Blood and buccal cells will be collected from donors to check for the presence of genotoxic permanent damage
Genotoxic evaluation by the Comet assay | Up to 1 year
  Blood will be analysed to check for the presence of genotoxic primary damage
Cytokine release | Up to 1 year
  Plasma will be analysed to check for the presence of cytokines
Microbiota analysis from feces by MinIOn | up to 1 year
  Feces will be analysed to check for variations in microbiota in the exposed and control groups

SECONDARY OUTCOMES:
Analyses of surrogate biomarkers | Up to 1 year
  Different metabolites will be analysed in the urine of participants, as an indirect measure to detect plastic exposure (p.eg. ftalates).
  The selection of the metabolite will depend of other analyses done on the project.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Catalan, Researcher, Principal Investigator — FIOH
Locations (4):
- Textile industry, Helsinki, Finland
- Spain (3):
  - Recycling company, Alicante
  - Textile Industry, Alicante
  - Control recruitment, Barcelona